CLINICAL TRIAL: NCT05949151
Title: Occlusal Forces and Muscle Activity in Fixed Versus Removable Mandibular Implant Supported Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asmaa Nabil Elboraey (Other)
Responsible Party: Sponsor-Investigator, Asmaa Nabil Elboraey, Associate Professor, National Research Centre, Egypt
Organization: National Research Centre, Egypt (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14312012023
Record Dates: First submitted 2023-06-30; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Occlusion
Keywords: implant supported overdenture; muscle activity
MeSH Terms: conditions — Bites and Stings | interventions — Dental Implants; Electromyography; Quality of Life

STUDY DESIGN:
Intervention Model Description: two group Group I: received a complete removable mandibular implant supported overdenture. While Group II: received implant supported fixed bridge.
Who Masked: Outcomes Assessor
Masking Description: the investigator didn't know which patients belonged to which group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Patients received a complete removable mandibular implant supported overdenture
  Interventions: Procedure: dental implants (K1 line conical connection double thread, OXY, Italy); Device: Occlusense (Bausch GmbH & Co. KG); Device: electromyography (EMG) (Nemus II)".; Other: oral health-related quality of life (OHRQoL)
- Group II (Active Comparator): Patients received implant supported fixed bridge
  Interventions: Procedure: dental implants (K1 line conical connection double thread, OXY, Italy); Device: Occlusense (Bausch GmbH & Co. KG); Device: electromyography (EMG) (Nemus II)".; Other: oral health-related quality of life (OHRQoL)

INTERVENTIONS:
Procedure: dental implants (K1 line conical connection double thread, OXY, Italy) — Six dental implants inserted on the edentulous mandible
Device: Occlusense (Bausch GmbH & Co. KG) — sensor used to evaluate the equilibration of occlusal forces.
Device: electromyography (EMG) (Nemus II)". — EMG recordings were accomplished by a computer electromyography-based data acquisition system
  Other Names: Assessment of Muscle Activity by electromyography (EMG) (Nemus II)
Other: oral health-related quality of life (OHRQoL) — Oral Health-related Quality of Life (OHRQoL) was estimated by employing the Oral Health Impact Profile questionnaire which comprises nineteen multiple questions that were translated into Arabic.

SUMMARY:
22 Patients having lower completely edentulous mandible aged 55-60 years were selected from the outpatient dental clinic of the Medical Excellence Centre of the National Research (NRC) Cairo, Egypt. Six dental implants were inserted in the mandible of each patient.

The patients were randomly categorized into two groups according to the final restoration.

DETAILED DESCRIPTION:
Group I: received a complete removable mandibular implant supported overdenture. While Group II: received implant supported fixed bridge.

Occlusal equilibrations, Muscle activities, and oral health-related quality of life (OHRQoL) were assessed by at the time of prosthesis insertion, after one and three month.

ELIGIBILITY:
Inclusion Criteria:

* edentulous mandible with well-developed alveolar ridge
* free from temporomandibular joint disorder
* free from any chronic diseases.

Exclusion Criteria:

* smoker
* patients having systemically immunosuppressive diseases
* patients receiving radiotherapy.

Ages: 55 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Occlusal equilibrations | Day 1 , one month and 3 month
  assessed by Occlusense device
Muscle activities | Day 1 , one month and 3 month
  assessed by Electromyograph (EMG) device

SECONDARY OUTCOMES:
oral health-related quality of life (OHRQoL) | Day 1, one month and 3 month
  Oral Health-related Quality of Life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Elboraey, Ass.Prof, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National Research Centre, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No